CLINICAL TRIAL: NCT05122442
Title: Multicenter, Non-interventional Study, Describing Patients With Inherited Retinal Disease (IRD) in France
Acronym: EPI-genRET
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8173
Record Dates: First submitted 2021-10-21; First posted 2021-11-16 (Actual); Results first posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-11

CONDITIONS: Inherited Retinal Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patients with inherited retinal disease — Patients with inherited retinal disease

SUMMARY:
Genetic diagnostic testing becomes increasingly important for enhancing our understanding of the disease notably the genetics and providing the best care to the patients, and several initiatives seek to gather more data in order to better understand and treat those diseases.

Within this context, Novartis and SENSGENE/Strasbourg University Hospitals (HUS) want to set up, through a research collaboration, a non-interventional study in France to better understand the epidemiology of IRDs, particularly the distribution of pathogenic variants in patients. This study aims to serve as a starter study to implement an IRD national registry led by SENSGENE/Strasbourg University Hospitals (HUS). The data collected might also be used to populate global European registries. The primary objective has been defined in a sufficient broad way to address this perspective of registries.

As IRDs can present from birth to late middle age, this study will include both children and adult patients regardless of age, sex, and the type of IRD.

ELIGIBILITY:
Inclusion criteria:

* All patients, whatever age or gender, clinically diagnosed with IRD or with high suspicion for IRDs based on clinical examination and functional tests (such as fundus exam and ERG), regardless of genetic testing
* Patients who attended a consultation at one of the participating centers from SENSGENE network over the inclusion period starting from sites initiation
* Patients who had been prescribed a genetic test for IRD prior to or at the date of inclusion.

Exclusion criteria:

* Patients/Parents/Legally authorized representatives (LAR) opposed to the collection and processing of their medical data/the medical data of their children/the medical data of the person for whom they are LAR;
* Patients who are suffering from any other retinal disorder or optic neuropathy that may clinically or genetically overlap with IRD or non-genetic (phenocopy);
* Patients/parents/Legally authorized representatives (LAR) refusing genetic testing;
* Patients lacking decision-making capacity: Mental incapacity, unwillingness, or language barriers precluding adequate understanding or cooperation.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with inherited retinal disease Attending a consultation in 7 IRD reference centres in France
Sampling Method: Probability Sample
Enrollment: 998 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Les Hôpitaux Universitaires, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Inherited Retinal Disease: All patients clinically diagnosed with IRD or with high suspicion for IRDs based on clinical examination and functional tests, regardless of genetic testing
Period: Overall Study
Arm/Group | Patients With Inherited Retinal Disease
Started | 998
Completed | 998
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 982 participants met study inclusion and exclusion criteria
Arm/Group | Patients With Inherited Retinal Disease
Number analyzed (Participants) | 982
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.92 (19.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 479
  Male | 503
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients by Type of IRD
Description: To describe the genetic testing characteristics To describe the distribution of variant of uncertain significance (VUS - class 3 variants) in IRD-associated genes To describe the proportion of unsolved patients To describe the type of pathogenic variants in each IRD-associated gene identified
Time Frame: 12 month
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Inherited Retinal Disease
Number analyzed (Participants) | 982
Participants
  Isolated progressive inherited retinal disorders | 720
  Syndromic inherited retinal disorders | 174
  Isolated stationary inherited retinal disorders | 30
  Other | 58

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Arm/Group | Patients With Inherited Retinal Disease
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/42/NCT05122442/Prot_SAP_000.pdf